CLINICAL TRIAL: NCT06899724
Title: A Randomized Multicentre Placebo Controlled Non-inferiority Study of Intravenous Sedation Versus Methoxyflurane During Hysteroscopy.
Brief Title: Methoxyflurane for Analgesia During Hysteroscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. John A. Thiel Medical Professional Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JThiel2
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Anesthetics, Inhalation; Methoxyflurane; Analgesia

STUDY DESIGN:
Intervention Model Description: Randomized double blind placebo controlled non-inferiority study
Who Masked: Participant, Care Provider, Investigator
Masking Description: After the interventions are assigned, an unblinded nurse will prepare the study medications according to each participant's identification number and treatment allocation group. Nursing staff in these clinics would normally prepare procedural medications. The nurse will prepare identical syringes filled with either fentanyl, midazolam, or normal saline, label the syringes with the participant identification number, and deliver them to the procedure room at the time of the scheduled hysteroscopy, confirming the patient's identity with the procedure team. They will also provide the Green Whistle and a vial of the methoxyflurane or saline. The physician, assisting nurses, and the participant will all be blinded to the identity of the medication in the syringe and the green whistle.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- IV Sedation (Active Comparator): Patients will receive 1 microgram/kg fentanyl and 1 - 3 mg midazolam intravenously as per the normal intravenous sedation protocol
  Interventions: Drug: Intravenous Sedatives with or Without Analgesia
- Methoxyflurane (Active Comparator): Patients will receive three inhalations from the green whistle loaded with methoxyflurane
  Interventions: Drug: Anesthetics, Inhalation
- IV saline (Placebo Comparator): Patients in the Methoxyflurane group will receive intravenous saline administered from the same syringes as those in the fentanyl and midazolam group
  Interventions: Drug: Anesthetics, Inhalation
- Inhaled saline (Placebo Comparator): Patients in the Intravenous sedation group will receive three inhalations of saline from a placebo loaded green whistle
  Interventions: Drug: Intravenous Sedatives with or Without Analgesia

INTERVENTIONS:
Drug: Anesthetics, Inhalation — Inhaled analgesia
  Other Names: Methoxyflurane
  Arms: IV saline; Methoxyflurane
Drug: Intravenous Sedatives with or Without Analgesia — IV Fentanyl and midazolam
  Arms: IV Sedation; Inhaled saline

SUMMARY:
This study is to assess the non-inferiority of using inhaled methoxyflurane (MOF) versus intravenous conscious sedation with fentanyl and midazolam on women's perception of pain, during hysteroscopy and/or polypectomy in an outpatient setting. The researchers will determine whether the participants receiving the inhaled MOF (experimental group) achieve similar clinical effects in reduction of pain and ability to complete the procedure. Women's perception of pain will be recorded on a scale from 0 to 10 using the numeric rating scale (NRS).

DETAILED DESCRIPTION:
Methoxyflurane (MOF) is a halogenated hydrocarbon volatile general anesthetic that was discontinued in the 1960s due to potential nephrotoxicity. It was subsequently found that at sub-anesthetic doses, it was safe, with no risk of renal impairment, and provided excellent procedural analgesia. The mechanism of action for the analgesic effect is unclear, although it may be related to an effect on substance P and beta-endorphin levels. It is indicated for use for the short-term relief of moderate to severe pain associated with procedures in adults and may be safely used in the geriatric population (>65 years). It has a rapid onset and short half-life, so the effects rapid resolve following procedures (1).

MOF is indicated for self-administration under the supervision of medical personnel for procedural pain and has been safely used in over 5 million patients (2). The use of MOF for procedural analgesia does not affect systemic blood pressure, respiratory rate, or consciousness (2, 3, 4). The most common adverse effects include dizziness, confusion, feeling intoxicated, nausea, and a bad taste. A number of studies have shown no serious adverse events during usage for various procedures (4, 5, 6, 7). It should be avoided in patients with significant renal disease, a history of impaired hepatic function after the use of halogenated anesthetic agents, malignant hyperthermia, and clinically evident hemodynamic or respiratory depression. It should also be avoided in patients using opiates, sedatives, hypnotics, phenothiazines, tranquilizers, skeletal muscle relaxants, alcohol, and potentially nephrotoxic medications.

MOF is self-administered under the supervision of a health care professional using an inhaler (green whistle) that is loaded with 3 cc of 99.9% methoxyflurane. The inhalation device includes an activated carbon chamber that absorbs the exhaled MOF to avoid anesthetic pollution of the procedure room (1). The effects of the medication on psychomotor function return to baseline levels when compared to placebo in a number of tests, including auditory reaction time, hand-eye coordination, and logical reasoning (8). This would allow the patient to return to highly skilled activities such as work or driving on the day of the procedure.

Hysteroscopy is one of the most commonly performed procedures in gynecology (9). Relocating gynecologic procedures such as hysteroscopy from the operating room to an ambulatory setting improves resource allocation and access to the OR for other patients while also improving the patient experience (9). In some centers, this move encounters a significant barrier in providing adequate analgesia. Ineffective analgesia can lead to incomplete or suboptimal assessment and management of pathology (10, 11). The large variance in analgesic options, ranging from oral non-steroidal anti-inflammatories or opiates to intravenous opiates, suggests that there is no single best option.

Sairally et al. (2024) reported that up to a third of patients undergoing hysteroscopy experience severe pain, which may result in procedures being completed in an operating room setting. This can be overcome with intravenous sedation rather than oral analgesia or nitrous oxide; however, access to nurse-administered intravenous (IV) sedation may be limited, and removing an anesthetist from the operating room limits case numbers that can be done there.

The current standard for ambulatory analgesia in most Canadian centers is intravenous sedation with fentanyl and midazolam. This is an effective option, but it requires intravenous access and monitoring of vital signs during and after the procedure. Both opiate and benzodiazepine medications have well-known potential risks, including hypotension, hypoxia, and somnolence. There is often a need for prolonged post-procedure monitoring, especially in the older age groups, which can limit the number of procedures completed in a given amount of time.

The use of inhaled methoxyflurane (Penthrox) has been shown to provide appropriate and effective analgesia for ambulatory care settings with less need for prolonged post-procedure monitoring with quicker recovery and discharge from care. Several studies have examined the effectiveness of methoxyflurane (MOF) use during orthopedic, general surgery, and urological day procedures and with brachytherapy (3, 7, 9, 12, 13, 14, 15, 16, 17). One recent study (9) demonstrated that the use of MOF during hysteroscopy and/or polypectomy and other ambulatory gynecologic procedures was effective, well tolerated with no serious adverse effects. Twidale et al (2022) noted that using MOF during hysteroscopy significantly reduced pain for patients compared to inhaled nitrous oxide.

Debuka et al (2023) showed that removal of orthopaedic external fixator hardware could be completed using methoxyflurane (MOF) rather than the usual general anesthetic or regional block. The average mean visual analogue score (VAS) was 3.9, and patient satisfaction with the level of analgesia was >95%. The authors estimated that relocating these procedures to an ambulatory setting freed up about 80 hours of operating room time a year in their center and reduced the cost per hour from 283 pounds to 24 pounds. The included ages of participants were 19 to 85 years of age, which would be comparable to those undergoing hysteroscopy.

Locke et al (2024) found that replacing intravesical lidocaine with inhaled MOF for cystoscopic procedures was efficacious, had high levels of patient satisfaction and was associated with a VAS score of 4 +/- SD 2.6. Elterman et al (2022) found that using MOF during rigid cystoscopy and water vapour therapy for benign prostatic enlargement in a population with a mean age of 72 resulted in VAS scores of zero. Stewart et al (2023) found that using MOF during cervical brachytherapy applicator removal significantly reduced median pain scores for both retrospective recall and prospective evaluation.

In a randomized, multicentre, non-blinded randomized control trial, Nguyen et al. (2013) compared IV fentanyl and midazolam versus MOF use during colonoscopies and noted no difference in VAS scores before, during, and after the procedure. The procedure preparation time, total time in the room, and procedure success (including polyp detection and removal) were no different between IV sedation and MOF. The MOF group had no reported oxygen desaturations, awoke quicker, and were ready for discharge sooner than the IV sedation group. Ninety-seven percent of the patients said they would use MOF again for colonoscopy.

Nguyen et al (2015) used the same protocol for colonoscopy on patients who were morbidly obese or had sleep apnea. The patients did report more pain in the MOF group but noted this pain was tolerable, and there was no difference in pain scores following the procedure. The preparation time, total time in the room, and procedural success were again similar in the two groups. The MOF group experienced less respiratory depression, hypotension, and tachycardia. This group had a shorter time to be fully awake and were ready for discharge sooner than the intravenous sedation group.

Hayne et al (2022) noted in a multicenter, randomized double-blind placebo-controlled trial in men undergoing their first TRUS-guided prostate biopsy that there were lower scores for pain (mean 2.51 MOF VS. 2.82 PLA; 95% CI -0.75-0.14; p=0.18) and an improved patient experience in the MOF group. There were no adverse events reported, and after 15 minutes, there was no difference in the discomfort in the two groups. Copping et al (2024), in a randomized double-blind placebo-controlled study, found that the use of MOF during portacath insertion and removal and solid organ biopsy resulted in reduced pain scores, lower patient anxiety, and no serious adverse events.

Spruyt et al (2014) completed a single site randomized double-blind placebo-controlled study for bone marrow biopsy showing significant reduction in the worst pain scores in the MOF group compared to placebo (3.3 ±2.0 vs 5.0 ±2.4, p<0.001) (17). The reported adverse events were minor, including dizziness, euphoria, and flushing. Significantly more patients rated the procedure experience as very good to excellent in the MOF group (63% vs 50%).

Although there is somewhat limited evidence for the use of MOF for procedural analgesia in the literature (21, 22), there are a number of quality studies that have demonstrated the safety and efficacy of MOF. There are no reported serious adverse events. The minor complications, including dizziness, nausea, flushing, and drowsiness, all resolve quickly. None of the trials reported hypotension, respiratory depression, or significant cardiac issues. Since MOF has been an effective analgesic for several ambulatory procedures, it has excellent potential to provide a safe, reproducible, and effective analgesia for ambulatory hysteroscopy and/or polypectomy.

References

1. Penthrox product monograph. Paladin Labs Inc, 100 Alexis-Nihon Blvd, Suite 600, St-Laurent, Quebec, Canada.
2. Jephcott, C, J Grummet, N. Nguyen, O. Spruyt. 2018. A review of the safety and efficacy of inhaled methoxyflurane as an analgesic for outpatient procedures. British Journal of Anaesthesia 120:1040-1048.
3. Debuka E, P Birkenhead, S Shah, B Narayan, N Giotakis, P Thorpe, SM Graham, BE Fischer, N Peterson. 2023. Penthrox (methoxyflurane) as an analgesic for removal of circular external fixators and minor procedures during the COVID-19 pandemic. Strategies in Trauma and Limb Reconstruction 18:82-86.
4. Trimmel H, A Egger, R Doppler, M Pimiskern, WG Voelckel. 2022. Usability and effectiveness of inhaled methoxyflurane for prehospital analgesia - a prospective, observational study. BMC Emergency Medicine 22:8-17.
5. Mercadante S, A. Voza, S Serra, F Ruggiano, F Carpinteri, G Gangitano, F Intelligente, E Bonafede, A Sblendido, A Farina, A Soldi, A Fabbri. 2019. Analgesic efficacy, practicality and safety of inhaled methoxyflurane versus standard analgesic treatment for acute trauma pain in the emergency setting: a randomised, open-label, active controlled, multicentre trial in Italy (MEDITA). 2019. Advanced Therapeutics 36:3030-3046.
6. Locke JA, S Neu, J Lawrence, S Herschorn. Pilot study to assess the feasibility of self-administered, low dose methoxyflurane for cystoscopic procedures. 2024. Canadian Urology Association Journal 18:251-254.
7. Nguyen NQ, L Toscano, M Lawrence, J Moore, RH Holloway, D Bartholomeusz, I Lidums, W Tam, IC Roberts-Thomson, VN Mahesh, TI Debreceni, MN Schoeman. 2013. Patient-controlled analgesia with inhaled methoxyflurane versus conventional endoscopist-provided sedation for colonoscopy: a randomized multicentre trial. Gastronintestinal Endoscopy 78:892-901.
8. Nguyen NQ, J Burgess, TL Debreceni, L Toscano. 2016. Psychomotor and cognitive effects of 15 minute inhalation of methoxyflurane in healthy volunteers: implication for post-colonoscopy care. Endoscopy International Open 04:E1171-1177
9. Sairally BZF, PP Smith, PM De Silva, S O'Connor, C Yates and TJ Clark. 2024. Inhaled methoxyflurane (Penthrox) as a novel pain relief for outpatient hysteroscopy and other gynaecological procedures. 2024. 302:206-210.
10. Ahmad G, Saluja S, O'Flynn H, Sorrentino A, Leach D, Watson A. 2017. Pain relief for outpatient hysteroscopy (Review). Cochrane Database of Systematic Reviews 10:1-80.
11. De Silva P, Mahmud A, Smith PP and Clark TJ. 2020. Analgesia for office hysteroscopy: A systematic revierw and meta-analysis. Journal of Minimally Invasive Gynecology 27:1034-1047.
12. Dias AV, Z Zeidan, M Copp, F Eslabra, R Hassan, R Middleton. 2024. Penthrox is an effective analgesia but is it patient approved? Cureus 16:e53537. DOI 10.7759/cureus.53537.
13. Smith MD, E Rowan, R Spaight, AN Siriwardena. 2022. Evaluation of the effectiveness and costs of inhaled methoxyflurane versus usual analgesia for prehospital injury and trauma: non-randomised clinical study. 2022. BMC Emergency Medicine 22:122-136.
14. Wong KY, JS Ki Lau, AY Chung Siu, PG Kan. A randomized non-inferiority pilot study on the use of methoxyflurane (Penthrox) for pain control in the emergency department. Hong Kong Journal of Emergency Medicine 29:203-211.
15. Elterman DS, KC Zorn, N Bhojani, B Chughtai. 2022. Efficacy and safety of methoxyflurane (Penthrox) for pain control during water vapor thermal therapy (Rezun) for benign prostatic enlargement. Canadian Journal of Urology 29:11355-11360.
16. Twidale EK, Neutens S, Hynt L, Dudley N, Streeton C. 2024. Methoxyflurane analgesia for outpatient hysteroscopy: a double-blind, randomised, controlled trial. Australian New Zealand Journal of Obstetrics and Gynecology DOI; 10.111/ajo.13861.
17. Stewart AJ, C Brookr, G Vose, K Redmond, A Williams, N Pankhania, H Dommett, J Kirk-Bayley, AP Franklin, B Morrison. 2023. Pain and symptom relief using inhaled methoxyflurane for gynecologic brachytherapy applicator removal. Journal of Contemporary Brachytherapy 15:37-42.
18. Hayne D, J Grummet, D Espinoza, SP McCombie, V Chalasani, KS Ford, M Frydenberg, P Gilling, B Goreon, C Hawks, A Konstantatos, AJ Martin, A Nixon, C O'Brien, MI Patel, S Sengupta, S Shahbaz, S Subramaniam, S Williams, HH Woo, MR Stockler, ID Davis, N Buchan. 2022. Pain-free TRUS B': a phase 3 double-blind placebo-controlled randomized trial lof methoxyflurane with periprostatic local anaesthesia to reduce the discomfort of transrectal ultrasonography-guided prostate biopsy (ANZUP 1501). BJU International 129:591-600.
19. Copping R, P Balamon, M Lau, J Catt, G Schlapoff. 2024. MethOxyfluraNe in InTerventional Radiology (MONITOR): a randomized controlled trial. 2024. Journal of Medical Imaging in Radiation Oncology 68:705-713.
20. Spruyt O, D Westerman, A Milner, M Bressel, S Wein. 2014. A randomised, double-blind, placebo-controlled study to assess the safety and efficacy of methoxyflurane for procedural pain of a bone marrow biopsy. BMJ Supportive and Palliative Care 4:343-348.
21. Methoxyflurane inhalation as an analgesic for minor gynecological, ambulatory or emergency procedures. 2024.n Canadian Agency for Drugs and Techologies in Health (CADTH) Rapid Review. Report No. RC1545, Ottawa, Ontario, Canada.
22. Coffey F, P Dissmann, K Mirza, M Lomax. Methoxyflurane analgesia in adult patients in the emergency department: a subgroup analysis of a randomized, double-blind, placebo-controlled study (STOP). 2016 33:2012-2031.

ELIGIBILITY:
Inclusion Criteria:

Abnormal uterine Bleeding requiring hysteroscopy Postmenopausal bleeding requiring hysteroscopy

Exclusion Criteria:

Uterine or patient characteristics that preclude hysteroscopy Submucosal fibroids requiring myomectomy Past allergic reaction to fentanyl or midazolam BMI > 42 Contraindications precluding use of intravenous sedation (sleep apnea) Lack of patient consent History of malignant hyperthermia History of significant renal or hepatic disease

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Patient analgesia | 15, 30 and 60 seconds
  Patients will rate their pain on a Numeric Rating Scale during the procedure

SECONDARY OUTCOMES:
Time to complete procedure | 15 minutes
  Time required from surgeon start to completion
Pain one hour post procedure | 60 minutes post procedure
  Patients will rate their pain on the Numeric Rating Scale
Rescue analgesia | 60 minutes
  Any need for rescue analgesia during or after the procedure will be recorded
Acceptability of the procedure | 60 minutes
  Patients will be asked to rate the acceptability of the procedure on the Numeric Rating Scale and if they would recommend the procedure to a friend
Time to discharge | 60 minutes
  The time from return to the recovery area to the patient meeting criteria to be safe for discharge will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Thiel, MD MPH FRCSC, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Penthrox product monograph. Paladin Labs Inc, 100 Alexis-Nihon Blvd, Suite 600, St-Laurent, Quebec, Canada.
- [Background] Jephcott C, Grummet J, Nguyen N, Spruyt O. A review of the safety and efficacy of inhaled methoxyflurane as an analgesic for outpatient procedures. Br J Anaesth. 2018 May;120(5):1040-1048. doi: 10.1016/j.bja.2018.01.011. Epub 2018 Feb 12. PMID 29661381
- [Background] Debuka E, Birkenhead P, Shah S, Narayan B, Giotakis N, Thorpe P, Graham SM, Fischer BE, Peterson N. Penthrox(R) (Methoxyflurane) as an Analgesic for Removal of Circular External Fixators and Minor Procedures during the COVID-19 Pandemic. Strategies Trauma Limb Reconstr. 2023 May-Aug;18(2):82-86. doi: 10.5005/jp-journals-10080-1587. PMID 37942432
- [Background] Trimmel H, Egger A, Doppler R, Pimiskern M, Voelckel WG. Usability and effectiveness of inhaled methoxyflurane for prehospital analgesia - a prospective, observational study. BMC Emerg Med. 2022 Jan 15;22(1):8. doi: 10.1186/s12873-021-00565-6. PMID 35033003
- [Background] Mercadante S, Voza A, Serra S, Ruggiano G, Carpinteri G, Gangitano G, Intelligente F, Bonafede E, Sblendido A, Farina A, Soldi A, Fabbri A; MEDITA Study Group. Analgesic Efficacy, Practicality and Safety of Inhaled Methoxyflurane Versus Standard Analgesic Treatment for Acute Trauma Pain in the Emergency Setting: A Randomised, Open-Label, Active-Controlled, Multicentre Trial in Italy (MEDITA). Adv Ther. 2019 Nov;36(11):3030-3046. doi: 10.1007/s12325-019-01055-9. Epub 2019 Oct 12. PMID 31612359
- [Background] Locke JA, Neu S, Lawrence J, Herschorn S. Pilot study to assess the feasibility of self-administered, low-dose methoxyflurane for cystoscopic procedures. Can Urol Assoc J. 2024 Aug;18(8):251-254. doi: 10.5489/cuaj.8676. PMID 38587974
- [Background] Nguyen NQ, Toscano L, Lawrence M, Moore J, Holloway RH, Bartholomeusz D, Lidums I, Tam W, Roberts-Thomson IC, Mahesh VN, Debreceni TL, Schoeman MN. Patient-controlled analgesia with inhaled methoxyflurane versus conventional endoscopist-provided sedation for colonoscopy: a randomized multicenter trial. Gastrointest Endosc. 2013 Dec;78(6):892-901. doi: 10.1016/j.gie.2013.05.023. Epub 2013 Jun 28. PMID 23810328
- [Background] Nguyen NQ, Burgess J, Debreceni TL, Toscano L. Psychomotor and cognitive effects of 15-minute inhalation of methoxyflurane in healthy volunteers: implication for post-colonoscopy care. Endosc Int Open. 2016 Nov;4(11):E1171-E1177. doi: 10.1055/s-0042-115409. Epub 2016 Nov 8. PMID 27853742
- [Background] Sairally BZF, Smith PP, De Silva PM, O'Connor S, Yates C, Clark TJ. Inhaled methoxyflurane (Penthrox(R)) as a novel pain relief for outpatient hysteroscopy and other gynaecological procedures. Eur J Obstet Gynecol Reprod Biol. 2024 Nov;302:206-210. doi: 10.1016/j.ejogrb.2024.09.002. Epub 2024 Sep 6. PMID 39303369
- [Background] Ahmad G, Saluja S, O'Flynn H, Sorrentino A, Leach D, Watson A. Pain relief for outpatient hysteroscopy. Cochrane Database Syst Rev. 2017 Oct 5;(10)(10):CD007710. doi: 10.1002/14651858.CD007710.pub3. PMID 35611933
- [Background] De Silva PM, Mahmud A, Smith PP, Clark TJ. Analgesia for Office Hysteroscopy: A Systematic Review and Meta-analysis. J Minim Invasive Gynecol. 2020 Jul-Aug;27(5):1034-1047. doi: 10.1016/j.jmig.2020.01.008. Epub 2020 Jan 23. PMID 31982584
- [Background] Dias AV, Zeidan Z, Copp M, Eslabra F, Hassan R, Middleton R. Penthrox Is an Effective Analgesic but Is It Patient Approved? Cureus. 2024 Feb 4;16(2):e53537. doi: 10.7759/cureus.53537. eCollection 2024 Feb. PMID 38445124
- [Background] Smith MD, Rowan E, Spaight R, Siriwardena AN. Evaluation of the effectiveness and costs of inhaled methoxyflurane versus usual analgesia for prehospital injury and trauma: non-randomised clinical study. BMC Emerg Med. 2022 Jul 7;22(1):122. doi: 10.1186/s12873-022-00664-y. PMID 35799131
- [Background] 14. Wong KY, JS Ki Lau, AY Chung Siu, PG Kan. A randomized non-inferiority pilot study on the use of methoxyflurane (Penthrox) for pain control in the emergency department. Hong Kong Journal of Emergency Medicine 29:203-211.
- [Background] Elterman DS, Zorn KC, Bhojani N, Chughtai B. Efficacy and safety of methoxyflurane (Penthrox) for pain control during water vapor thermal therapy (Rezum) for benign prostatic enlargement. Can J Urol. 2022 Dec;29(6):11355-11360. PMID 36495576
- [Background] Twidale EK, Neutens S, Hynt L, Dudley N, Streeton C. Methoxyflurane analgesia for outpatient hysteroscopy: A double-blind, randomised, controlled trial. Aust N Z J Obstet Gynaecol. 2025 Feb;65(1):69-76. doi: 10.1111/ajo.13861. Epub 2024 Jul 15. PMID 39007504
- [Background] Stewart AJ, Brooker C, Vose G, Redmond K, Williams A, Pankhania N, Dommett H, Kirk-Bayley J, Franklin AP, Morrison B. Pain and symptom relief using inhaled methoxyflurane for gynecologic brachytherapy applicator removal. J Contemp Brachytherapy. 2023 Feb;15(1):37-42. doi: 10.5114/jcb.2023.125581. Epub 2023 Feb 28. PMID 36970443
- [Background] Hayne D, Grummet J, Espinoza D, McCombie SP, Chalasani V, Ford KS, Frydenberg M, Gilling P, Gordon B, Hawks C, Konstantatos A, Martin AJ, Nixon A, O'Brien C, Patel MI, Sengupta S, Shahbaz S, Subramaniam S, Williams S, Woo HH, Stockler MR, Davis ID, Buchan N; Australian and New Zealand Urogenital and Prostate Cancer Trials Group (ANZUP). 'Pain-free TRUS B': a phase 3 double-blind placebo-controlled randomized trial of methoxyflurane with periprostatic local anaesthesia to reduce the discomfort of transrectal ultrasonography-guided prostate biopsy (ANZUP 1501). BJU Int. 2022 May;129(5):591-600. doi: 10.1111/bju.15552. Epub 2021 Jul 30. PMID 34273231
- [Background] Copping R, Balamon P, Lau M, Catt J, Schlaphoff G. MethOxyfluraNe in InTerventiOnal Radiology (MONITOR): A randomised controlled trial. J Med Imaging Radiat Oncol. 2024 Sep;68(6):705-713. doi: 10.1111/1754-9485.13726. Epub 2024 Jun 25. PMID 38923825
- [Background] Spruyt O, Westerman D, Milner A, Bressel M, Wein S. A randomised, double-blind, placebo-controlled study to assess the safety and efficacy of methoxyflurane for procedural pain of a bone marrow biopsy. BMJ Support Palliat Care. 2014 Dec;4(4):342-8. doi: 10.1136/bmjspcare-2013-000447. Epub 2013 Jun 7. PMID 24644183
- [Background] Methoxyflurane Inhalation as an Analgesic for Minor Gynecological, Ambulatory, or Emergency Procedures: Rapid Review [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2024 Sep. Report No.: RC1545. Available from http://www.ncbi.nlm.nih.gov/books/NBK608473/ PMID 39466939
- [Background] Coffey F, Dissmann P, Mirza K, Lomax M. Methoxyflurane Analgesia in Adult Patients in the Emergency Department: A Subgroup Analysis of a Randomized, Double-blind, Placebo-controlled Study (STOP!). Adv Ther. 2016 Nov;33(11):2012-2031. doi: 10.1007/s12325-016-0405-7. Epub 2016 Aug 27. PMID 27567918
- [Background] 23. Sealed Envelope Ltd. 2012. Power calculator for continuous outcome non-inferiority trial. [Online] Available from: https://www.sealedenvelope.com/power/continuous-noninferior/ [Accessed Wed Feb 05 2025].